CLINICAL TRIAL: NCT04013152
Title: French Prospective Clinical Database of Colorectal Robotic Surgery
Brief Title: Clinical Database of Colorectal Robotic Surgery
Acronym: ROBOT CR
Status: Active, not recruiting | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: PROICM 2017-05 ROB
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease; Polyposis; Ulcerative Colitis; Diverticulitis; Colorectal Tumor; Rectal Prolapse; Benign Colorectal Tumor
Keywords: CROHN; Diverticulitis; Rectal; colorectal; ulcerative; colitis; polyposis; rectum; prolapse
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Diverticulitis; Colorectal Neoplasms; Rectal Prolapse; Ulcer; Colitis; Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- clinical database
  Interventions: Other: Clinical database

INTERVENTIONS:
Other: Clinical database — Constitution of a prospective, multicenter clinical database of surgery with robotic assistance in colorectal pathologies

SUMMARY:
Evaluation of robot Da Vinci Xi by determining its learning curve.The operating time will be defined by patient then the operating average will be calculated.

DETAILED DESCRIPTION:
Since the emergence of minimally invasive technology twenty years ago, as a surgical concept and surgical technique for colorectal cancer surgery, its obvious advantages have been recognized.

Laparoscopic technology, as one of the most important technology platform, has got a lot of evidence-based support for the oncological safety and effectiveness in colorectal cancer surgery Laparoscopic technique has advantages in terms of identification of anatomic plane and autonomic nerve, protection of pelvic structure, and fine dissection of vessels.

But because of the limitation of laparoscopic technology there are still some deficiencies and shortcomings, including lack of touch and lack of stereo vision problems, in addition to the low rectal cancer, especially male, obese, narrow pelvis, larger tumors, it is difficult to get better view and manipulating triangle in laparoscopy. However, the emergence of a series of new minimally invasive technology platform is to make up for the defects and deficiencies. The robotic surgical system possesses advantages, such as stereo vision, higher magnification, manipulator wrist with high freedom degree, filtering of tremor and higher stability, but still has disadvantages, such as lack of haptic feedback, longer operation time, high operation cost and expensive price.

3D system of laparoscopic surgery has similar visual experience and feelings as robotic surgery in the 3D view, the same operating skills as 2D laparoscopy and a short learning curve. Transanal total mesorectal excision (taTME) by changing the traditional laparoscopic pelvic surgery approach, may have certain advantages for male cases with narrow pelvic and patients with large tumor.

No prospective study has compared these four surgical techniques. Furthermore, the learning curve still remains a crucial problem in term of data interpretation.

We will collect synchronized videos and data on surgeon performance during colorectal surgeries using the Vinci Logger (dVLogger, Intuitive Surgical, Inc.), it is a personalized recording tool that captures synchronized video in the form of endoscope view at 30 frames per second. Kinematic data included characteristics of movement such as instrument travel time, path length and velocity. Events included frequency of master controller clutch use, camera movements, third arm swap and energy use.

We will explore and validate objective surgeon performance metrics using novel recorder ("dVLogger") to directly capture surgeon manipulations on the daVinci Surgical System.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Colorectal pathologies (Crohn's disease, Polyposis, Ulcerative colitis, Diverticulitis, Colorectal tumor, Rectal prolapse, Benign and colorectal tumor) eligible for robotic surgery.
3. Major techniques: right and left colectomy, rectal excision (low anterior resection, intersphincteric resection, abdominoperineal resection), Hartman reversal
4. Or, Minor techniques: rectopexy, shaving for rectal endometriosis,
5. Or, Complex techniques: extended rectal excision for T4 cancer, pelvectomy, redo surgery.
6. Patient affiliated to a social security regimen
7. Patient information for study

Exclusion Criteria:

1. Legal incapacity or physical, psychological social or geographical status interfering with the patient's ability to agree to participate in the study
2. Patient under tutelage, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal tumor, Crohn's disease, Polyposis, Ulcerative colitis, Diverticulitis, Rectal prolapse, Benign colorectal tumor
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2027-06-09 (Estimated)

PRIMARY OUTCOMES:
Collection of clinical data following surgery with robotic assistance in colorectal pathologies | 3 years

SECONDARY OUTCOMES:
Time of learning for each surgical technique by determining a learning curve for each of them | 3 years
The conversion rate of surgical technique | 3 years
Operating time | 3 years
Intraoperative complications rate | 3 years
Duration of hospital stay | 1 month
local relapse-free survival | 8 years
overall survival | 8 years
Digestive functionality assessment by using the Low Anterior Resection Syndrome score (LARS) | 3 years
  This questionnaire assessed the bowel function of patient. The range is from 8 (low function) to 35 (high function)
The Erectile Function of patient by using the II-EF-5 score (The International Index of Erectile Function) | 3 years
  The range is from 1 (low erectile function) to 27 (high erectile function)
The dysfunction of female Sexual Function by using the Index FSFI (The Female Sexual Function Index) score | 3 years
  The range is from 3 (low sexual function) to 55 (high sexual function).
Urinary functionality by using the questionnaire of urinary function | 3 years
  The range is from 0 (low urinary function) to 40 (high urinary function).
Objective surgeon performance metrics using a novel recorder (dVLogger) to directly capture surgeon manipulations on the da Vinci Surgical System | 3 years
Number of lymph node resected | 3 years
Quality of the mesorectum by using Quirke classification | 3 years
  The quality of the mesorectum resection is determined by the pathologist according to the aspect of mesorectum, the circumferential resection margin, cone effect .

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rouanet, MD, Study Chair — Institut régional du cancer de Montpellier
Locations (4):
- France (4):
  - CHU de Bordeaux, Bordeaux, Gironde
  - Institut régional du cancer de Montpellier, Montpellier, Hérault
  - CHU de Clermont-Ferrand, Clermont-Ferrand, Puy De Dôme
  - CHU de Lyon, Lyon, Rhône

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colombo PE, Bertrand MM, Alline M, Boulay E, Mourregot A, Carrere S, Quenet F, Jarlier M, Rouanet P. Robotic Versus Laparoscopic Total Mesorectal Excision (TME) for Sphincter-Saving Surgery: Is There Any Difference in the Transanal TME Rectal Approach? : A Single-Center Series of 120 Consecutive Patients. Ann Surg Oncol. 2016 May;23(5):1594-600. doi: 10.1245/s10434-015-5048-4. Epub 2015 Dec 29. PMID 26714950
- [Background] Bertrand MM, Colombo PE, Mourregot A, Traore D, Carrere S, Quenet F, Rouanet P. Standardized single docking, four arms and fully robotic proctectomy for rectal cancer: the key points are the ports and arms placement. J Robot Surg. 2016 Jun;10(2):171-4. doi: 10.1007/s11701-015-0551-y. Epub 2015 Dec 8. PMID 26645073
- [Background] Nagtegaal ID, van de Velde CJ, van der Worp E, Kapiteijn E, Quirke P, van Krieken JH; Cooperative Clinical Investigators of the Dutch Colorectal Cancer Group. Macroscopic evaluation of rectal cancer resection specimen: clinical significance of the pathologist in quality control. J Clin Oncol. 2002 Apr 1;20(7):1729-34. doi: 10.1200/JCO.2002.07.010. PMID 11919228
- [Background] Chen SL, Steele SR, Eberhardt J, Zhu K, Bilchik A, Stojadinovic A. Lymph node ratio as a quality and prognostic indicator in stage III colon cancer. Ann Surg. 2011 Jan;253(1):82-7. doi: 10.1097/SLA.0b013e3181ffa780. PMID 21135690
- [Background] Zhang X, Wei Z, Bie M, Peng X, Chen C. Robot-assisted versus laparoscopic-assisted surgery for colorectal cancer: a meta-analysis. Surg Endosc. 2016 Dec;30(12):5601-5614. doi: 10.1007/s00464-016-4892-z. Epub 2016 Jul 11. PMID 27402096
- [Background] Parc Y, Reboul-Marty J, Lefevre JH, Shields C, Chafai N, Tiret E. Factors influencing mortality and morbidity following colorectal resection in France. Analysis of a national database (2009-2011). Colorectal Dis. 2016 Feb;18(2):205-13. doi: 10.1111/codi.13099. PMID 26299627
- [Background] Bege T, Lelong B, Esterni B, Turrini O, Guiramand J, Francon D, Mokart D, Houvenaeghel G, Giovannini M, Delpero JR. The learning curve for the laparoscopic approach to conservative mesorectal excision for rectal cancer: lessons drawn from a single institution's experience. Ann Surg. 2010 Feb;251(2):249-53. doi: 10.1097/SLA.0b013e3181b7fdb0. PMID 20040854
- [Background] Poloniecki J, Valencia O, Littlejohns P. Cumulative risk adjusted mortality chart for detecting changes in death rate: observational study of heart surgery. BMJ. 1998 Jun 6;316(7146):1697-700. doi: 10.1136/bmj.316.7146.1697. PMID 9614015
- [Background] Guend H, Widmar M, Patel S, Nash GM, Paty PB, Guillem JG, Temple LK, Garcia-Aguilar J, Weiser MR. Developing a robotic colorectal cancer surgery program: understanding institutional and individual learning curves. Surg Endosc. 2017 Jul;31(7):2820-2828. doi: 10.1007/s00464-016-5292-0. Epub 2016 Nov 4. PMID 27815742
- [Background] Bokhari MB, Patel CB, Ramos-Valadez DI, Ragupathi M, Haas EM. Learning curve for robotic-assisted laparoscopic colorectal surgery. Surg Endosc. 2011 Mar;25(3):855-60. doi: 10.1007/s00464-010-1281-x. Epub 2010 Aug 24. PMID 20734081
- [Background] Bolsin S, Colson M. The use of the Cusum technique in the assessment of trainee competence in new procedures. Int J Qual Health Care. 2000 Oct;12(5):433-8. doi: 10.1093/intqhc/12.5.433. PMID 11079224